CLINICAL TRIAL: NCT02903966
Title: A Multicentre, Randomised, Double-blind (Sponsor Unblinded), Placebo-controlled Study With Open Label Extension to Investigate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of GSK2982772 in Subjects With Active Ulcerative Colitis
Brief Title: GSK2982772 Study in Subjects With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202152; 2016-001833-29 (EudraCT Number)
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-04

CONDITIONS: Colitis, Ulcerative
Keywords: Tolerability; GSK2982772; Safety; Pharmacokinetics; RIP1 kinase inhibitor; Ulcerative colitis; Pharmacodynamics
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GSK2982772

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK2982772 in Part A double-blind phase (Experimental): Subjects will receive GSK2982772 60 mg orally three times daily (approximately 8 hours apart) for 42 days (6 weeks).
  Interventions: Drug: GSK2982772
- Placebo in Part A double-blind phase (Placebo Comparator): Subjects will receive placebo orally three times daily (approximately 8 hours apart) for 42 days (6 weeks).
  Interventions: Drug: Placebo
- GSK2982772 in Part B open label extension phase (Experimental): Subjects from GSK2982772 and placebo arm who complete Part A study will move to Part B open-label extension phase. All subjects will receive GSK2982772 60 mg three times daily (approximately 8 hours apart) for 42 days (6 weeks).
  Interventions: Drug: GSK2982772

INTERVENTIONS:
Drug: GSK2982772 — GSK2982772 is available as a 30 mg white to almost white, round film coated tablet which will be administered as two tablets three times a day as directed.
  Arms: GSK2982772 in Part A double-blind phase; GSK2982772 in Part B open label extension phase
Drug: Placebo — Placebo is available as a white to almost white, round film coated tablet which will be administered as two tablets three times a day as directed.
  Arms: Placebo in Part A double-blind phase

SUMMARY:
This study is the first experience with GSK2982772, a receptor-interacting protein-1 (RIP1) kinase inhibitor, in subjects with active ulcerative colitis (UC). The primary objective will be to investigate the safety and tolerability of repeat oral doses of GSK2982772 60 mg or placebo three times daily for 42 days (Part A) followed by open label with GSK298772 60 mg three times daily for 42 days (Part B). In addition to pharmacokinetics (PK), a number of experimental and clinical endpoints will be employed to obtain information on the pharmacodynamics (PD), and preliminary efficacy in subjects with active UC. Although no formal hypothesis will be tested, these endpoints will enable a broader understanding of the mechanism of action and potential for clinical efficacy of GSK2982772 in UC. Within 30 Days of screening visit, subjects will be randomized to receive either GSK2982772 60 mg or placebo orally three times daily for 42 Days (6 weeks) in a 2:1 ratio in Part A study. Subjects who complete the Part A study will move to open label Part B study to receive GSK2982772 60 mg three times daily for an additional 42 Days (6 weeks). After the open label (Part B) treatment period, subjects will enter the Follow-up period which lasts for 28 Days (+/- 3 Days) post the last administration of study medication. The total duration of participation in the study will be approximately 20 Weeks from screening to the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Subjects that do not have any medical conditions, other than active UC, that in the opinion of the Investigator put the subject at unacceptable risk or interfere with study assessments or integrity of the data. These medical conditions should be stable at the time of screening and are expected to remain stable for the duration of the study.
* Subject has had a confirmed diagnosis of active UC, as documented by complete diagnostic colonoscopy to the terminal ileum (TI) with biopsy performed >=3 months prior to screening. If diagnostic colonoscopy was not performed to the TI, it must be documented by the principal investigator that the subject has diffuse inflammation from the rectum extending proximally to the colon in a continuous and uniform way.
* A Complete Mayo Score of >=3 points and endoscopy sub score of 2 to 3 at screening, despite concurrent treatment with at least 1 of the following (oral corticosteroids or any oral 5-aminosalicylates (5-ASA) or purine analogues or all as defined): Oral 5-ASA at a stable dose (equivalent to >=2.4 grams per day (g/day) of Asacol) for at least 4 weeks prior to first dose. Must remain on a stable dose until end of treatment; Purine analogues (azathioprine, mercaptopurine, thiopurines) or methotrexate for at least 12 weeks prior to first dose. Must remain on a stable dose until end of treatment; Stable low dose oral corticosteroid (up to 20 mg prednisolone or equivalent) for 2 weeks prior to sigmoidoscopy. Must remain on a stable dose until end of treatment.
* If on rectal 5-ASA or corticosteroids, must remain on a stable dose for at least 4 weeks prior to first dose. Must remain on stable dose until the end of treatment.
* Subject is naive to any biological therapies for UC OR Subject may have had previous exposure to a single anti-tumor necrosis factor (TNF) biologic agent which was discontinued for reasons other than primary non-response more than 8 weeks (or 5 half-lives whichever is longer) prior to first dose OR Subject may have had previous exposure to a single biologic agent (example, vedolizumab) in the context of a previous clinical trial. The biologic agent must have been discontinued more than 8 weeks (or 5 half-lives whichever is longer) prior to first dose. Note: Exposure to a single biologic agent is not required in addition to inclusion criteria listed above (number fourth and fifth on the list).
* A body mass index (BMI) within range of 18.5 to 35 kilogram per meter square (kg/m^2) (inclusive) at screening.
* Male and Female subjects:

Males: Male subjects with female partners of child bearing potential must comply with the contraception requirements.

Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as 1) Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy. 2) Postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until at least 2 days after the last dose of study medication and completion of the follow-up visit. The Investigator is responsible for ensuring that subjects understand how to properly use methods of contraception.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and protocol.

Exclusion Criteria:

* Subject with diagnosis of indeterminate colitis, Crohn's Disease, infectious colitis, or ischemic colitis.
* Subject with fulminant UC, or UC limited to the rectum (disease extent <15 centimeters (cm) from the anal verge).
* Subject with previous small bowel or colonic surgery(with exception of appendectomy), histological evidence of colonic dysplasia or bowel stricture.
* Subject with colostomy, fistulae or known symptomatic stenosis of the intestine.
* Subject with toxic megacolon.
* Subject with positive Clostridium difficile toxin test or active/previous colonic cytomegalo virus (CMV) infection.
* Subject with current history of suicidal ideation behavior (SIB) as measures using the Columbia Suicide Severity Rating Scale (C-SSRS) or history of attempted suicide.
* An active infection, or a history of infections as follows:

Hospitalization for treatment of infection within 60 days before first dose (Day 1).

Currently on any suppressive therapy for a chronic infection (such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).

Use of parenteral (intravenous (IV) or intramuscular) antibiotics (antibacterials, antivirals, antifungals, or antiparasitic agents) for an infection within 60 days before first dose.

A history of opportunistic infections within 1 year of screening (example: pneumocystis jirovecii, CMV pnemonitis, aspergillosis). This does not include infections that may occur in immunocompetent individuals, such as fungal nail infections or vaginal candidiasis, unless it is of an unusual severity or recurrent nature.

Recurrent or chronic infection or other active infection that, in the opinion of the Investigator might cause this study to be detrimental to the patient.

History of tuberculosis (TB), irrespective of treatment status. A positive diagnostic TB test at screening defined as a positive QuantiFERON-TB Gold test or T-spot test. In cases where the QuantiFERON or T-spot test is indeterminate, the subject may have the test repeated once, but they will not be eligible for the study unless the second test is negative. In cases where the QuantiFERON or T-spot test is positive, but a follow-up chest x-ray, locally read by a radiologist, shows no evidence of current or previous pulmonary tuberculosis, the subject may be eligible for the study at the discretion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor.

* QTc >450 millisecond (msec) or QTc >480 msec for subjects with bundle branch block at screening.
* ALT >2 times upper limit of normal (ULN) and bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent) at screening.
* Current active or chronic history of liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Current or history of renal disease or estimated glomerular filtration rate (GFR) by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) calculation <60 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) at screening.
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency unless subject has a documented history of selective immunoglobulin A (IgA) deficiency.
* A major organ transplant (example: heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Any planned surgical procedure during the study.
* A history of malignant neoplasm within the last 5 years, except for adequately treated non-metastatic cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix that has been fully treated and shows no evidence of recurrence.
* The subject has received treatment with the protocol listed prohibited therapies or changes to those treatments, within the prescribed timeframe.

Other medications (including vitamins, herbal and dietary supplements) will be considered on a case-by-case basis, and will be allowed if in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.

* History of alcohol or drug abuse that would interfere with the ability to comply with the study.
* History of sensitivity to any of the study treatments, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Received a live or attenuated vaccine within 30 days of randomization OR plan to receive a vaccination during the study until 5 half-lives (or 2 days) plus 30 days after receiving GSK2982772.
* The subject has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer before the first dose of study medication, or plans to take part in another clinical trial (not inclusive of any UC registry study where no study medication is being administered) at the same time as participating in this clinical trial.
* Hemoglobin <10 grams per deciliter (g/dL); hematocrit <30 percent, white blood cell count <=3,000 per millimeter cube (mm^3) (<=3.0 into 10^9 per liter); platelet count <=100,000 per microliter (<=100 into 10^9 per liter); absolute neutrophil count <=1.5 into 10^9 per liter.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. As potential for and magnitude of immunosuppression with this compound is unknown, subjects with presence of hepatitis B core antibody (HBcAb) should be excluded.
* A positive serology for human immunodeficiency virus (HIV) 1 or 2 at screening.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (6):
  - GSK Investigational Site, Moreno Valley, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Marrero, Louisiana
  - GSK Investigational Site, Chesterfield, Michigan
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Cedar Park, Texas
- GSK Investigational Site, Ulm, Baden-Wurttemberg, Germany
- GSK Investigational Site, Amsterdam, Netherlands
- Poland (3):
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Ksawerów
  - GSK Investigational Site, Wroclaw
- Russia (6):
  - GSK Investigational Site, Kaliningrad
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Saint Pertersburg
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Ufa
- Sweden (2):
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- United Kingdom (3):
  - GSK Investigational Site, Stockport, Cheshire
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Dudley

REFERENCES:
- [Derived] Weisel K, Scott N, Berger S, Wang S, Brown K, Powell M, Broer M, Watts C, Tompson DJ, Burriss SW, Hawkins S, Abbott-Banner K, Tak PP. A randomised, placebo-controlled study of RIPK1 inhibitor GSK2982772 in patients with active ulcerative colitis. BMJ Open Gastroenterol. 2021 Aug;8(1):e000680. doi: 10.1136/bmjgast-2021-000680. PMID 34389633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the safety and tolerability of repeat oral doses of GSK2982772 60 milligram (mg) or placebo three times daily (TID) in Part A (double blind [DB]) followed by GSK2982772 60 mg TID in Part B open label extension (OL) in active ulcerative colitis (UC) participants.
Pre-assignment Details: A total of 77 participants were screened, of which 36 eligible participants were enrolled (41 were screening failure). All 36 participants were randomized to receive GSK2982772 60 mg or Placebo in Part A of the study.
Groups:
- Placebo TID DB /GSK2982772 60 mg TID OL: Eligible participants with UC, received two tablets of placebo TID orally for 42 days (from Day 1 to 43) in Part A (double blind phase), followed by GSK2982772 60 mg (given as 2 tablets of 30 mg) TID orally for 42 days (from Day 44 to 85) in Part B (open label phase). There was no wash out period in between Part A and B. All participants were followed up until Day 112.
- GSK2982772 60 mg TID DB/ GSK2982772 60 mg TID OL: Eligible participants with UC, received GSK2982772 60 mg (given as 2 tablets of 30 mg) TID orally for 42 days (from Day 1 to 43) in Part A (double blind phase), followed by GSK2982772 60 mg (given as 2 tablets of 30 mg) TID orally for 42 days (from Day 44 to 85) in Part B (open label phase). There was no wash out period in between Part A and B. All participants were followed up until Day 112. 1 participant was randomized to receive BID regimen instead of TID regimen prior to protocol amendment; however, BID and TID are presented in the same arm because the pharmacokinetic (PK) profile is comparable for BID & TID regimen.
Period: Part A (Day 1 to 43)
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB/ GSK2982772 60 mg TID OL
Started | 12 | 24
Completed | 11 | 24
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Part B (Day 44 to 112)
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB/ GSK2982772 60 mg TID OL
Started | 11 | 24
Completed | 11 | 22
Not Completed | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB/ GSK2982772 60 mg TID OL | Total
Number analyzed (Participants) | 12 | 24 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (11.17) | 39.0 (13.69) | 42.8 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 16 | 22
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  White - Arabic/North African Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 12 | 23 | 35

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Common (>=5%) Non-serious Adverse Events (Non-SAEs) and Any Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; other important medical events; is associated with liver injury and impaired liver function.
Time Frame: Up to Day 43
Population: Safety population comprised of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Placebo TID DB: Eligible participants with UC, received two tablets of placebo TID orally for 42 days in Part A (double blind phase).
- Part A: GSK2982772 60 mg TID DB: Eligible participants with UC, received GSK2982772 60 mg (given as 2 tablets of 30 mg) TID orally for 42 days in Part A (double blind phase).
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 12 | 24
Participants
  Common non-SAEs | 7 | 13
  Any SAEs | 1 | 0

2. Primary Outcome: Part B: Number of Participants With Common (>=5%) Non Serious AEs and SAEs
Description: as for outcome 1
Time Frame: From Day 44 to Day 112
Population: Safety Population. Only those participants with data available at the specified time points were analyzed. All participants in Part B were presented in a single arm as they all received GSK2982772 60 mg in Part B (OL Phase).
Measure: Count of Participants; unit: Participants
Groups:
- Part B: GSK2982772 60 mg TID OL: Eligible participants with UC, received GSK2982772 60 mg (given as 2 tablets of 30 mg) TID orally for 42 days in Part B (open label phase).
Arm/Group | Part B: GSK2982772 60 mg TID OL
Number analyzed (Participants) | 35
Participants
  Common non-SAEs | 7
  Any SAEs | 2

3. Primary Outcome: Part A: Number of Participants With Worst Case Abnormal Clinical Chemistry Parameters by Potential Clinical Importance (PCI) Criteria
Description: Clinical chemistry parameters with PCI ranges: aspartate amino transferase (AST), alanine amino transferase (ALT), and alkaline phosphatase (ALP) (high: >=2 times upper limit of normal [ULN] units per liter [U/L]); calcium (low: <2 millimoles per liter [mmol/L] and high: >2.75 mmol/L); glucose (low: <3 and high: >9 mmol/L); potassium (low: <3 and high: >5.5 mmol/L); sodium (low: <130 and high: >150 mmol/L); total bilirubin (high: >=1.5 times ULN micromoles per liter [µmol/L]); high density lipoproteins (HDL) 0.9 to 99.99 mmol/L; low density lipoprotein (LDL) 0 to 3.35 mmol/L; triglycerides 0 to 2.24 mmol/L, creatinine (high: change from Baseline [BL]>44.2 µmol/L). Participants were counted in the worst case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change'
Time Frame: Up to Day 43
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 12 | 24
Participants
  AST, To Low | 0 | 0
  AST, To within range or no change | 12 | 24
  AST, To High | 0 | 0
  ALT, To Low | 0 | 0
  ALT, To within range or no change | 12 | 24
  ALT, To High | 0 | 0
  ALP, To Low | 0 | 0
  ALP, To within range or no change | 12 | 24
  ALP, To High | 0 | 0
  Calcium, To Low | 0 | 0
  Calcium, To within range or no change | 12 | 24
  Calcium, To High | 0 | 0
  Glucose, To Low | 0 | 1
  Glucose, To within range or no change | 11 | 23
  Glucose, To High | 1 | 0
  Potassium, To Low | 0 | 0
  Potassium, To within range or no change | 12 | 24
  Potassium, To High | 0 | 0
  Sodium, To Low | 0 | 0
  Sodium, To within range or no change | 12 | 24
  Sodium, To High | 0 | 0
  Total Bilirubin, To Low | 0 | 0
  Total Bilirubin, To within range or no change | 12 | 24
  Total Bilirubin, To High | 0 | 0
  HDL, To Low | 0 | 0
  HDL, To within range or no change | 12 | 24
  HDL, To High | 0 | 0
  LDL, To Low | 0 | 0
  LDL, To within range or no change | 10 | 22
  LDL To High | 2 | 2
  Triglycerides, To Low | 0 | 0
  Triglycerides, To within range or no change | 12 | 23
  Triglycerides, To High | 0 | 1
  Creatinine, To Low | 0 | 0
  Creatinine, To within range or no change | 12 | 24
  Creatinine, To High | 0 | 0

4. Primary Outcome: Part B: Number of Participants With Worst Case Abnormal Clinical Chemistry Parameters by Potential Clinical Importance (PCI) Criteria
Description: Clinical chemistry parameters with their PCI ranges were: AST, ALT, and ALP (high: >=2 ULN [U/L]); calcium (low: <2 mmol/L and high: >2.75 mmol/L); glucose (low: <3 and high: >9 mmol/L); potassium (low: <3 and high: >5.5 mmol/L); sodium (low: <130 and high: >150 mmol/L); total bilirubin (high: >=1.5 times ULN [µmol/L]); HDL 0.9 to 99.99 mmol/L; LDL 0.to 3.35 mmol/L; triglycerides 0 to 2.24 mmol/L, creatinine (high: change from BL >44.2 µmol/L). Participants were counted in the worst case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: From Day 44 to Day 112
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK2982772 60 mg TID OL
Number analyzed (Participants) | 35
Participants
  AST, To Low | 0
  AST, To within range or no change | 35
  AST, To High | 0
  ALT, To Low | 0
  ALT, To within range or no change | 35
  ALT, To High | 0
  ALP, To Low | 0
  ALP, To within range or no change | 35
  ALP, To High | 0
  Calcium, To Low | 0
  Calcium, To within range or no change | 35
  Calcium, To High | 0
  Glucose, To Low | 1
  Glucose, To within range or no change | 34
  Glucose, To High | 0
  Potassium, To Low | 0
  Potassium, To within range or no change | 33
  Potassium, To High | 2
  Sodium, To Low | 0
  Sodium, To within range or no change | 35
  Sodium, To High | 0
  Total Bilirubin, To Low | 0
  Total Bilirubin, To within range or no change | 34
  Total Bilirubin, To High | 1
  HDL, To Low | 2
  HDL, To within range or no change | 33
  HDL, To High | 0
  LDL, To Low | 0
  LDL, To within range or no change | 33
  LDL, To High | 2
  Triglycerides, To Low | 0
  Triglycerides, To within range or no change | 34
  Triglycerides, To High | 1
  Creatinine, To Low | 0
  Creatinine, To within range or no change | 35
  Creatinine, To High | 0

5. Primary Outcome: Part A: Number of Participants With Worst Case Abnormal Hematology Parameters by PCI Criteria
Description: Hematology parameters with their PCI ranges were: hematocrit (high: >0.54 proportion of red blood cells in blood and low: change from BL<0.075); hemoglobin (high: >180 grams per liter [g/L] and low: change from BL<25 g/L); lymphocytes (low: <0.8 Giga cells/L); platelet count (low: <100 Giga cells/L and high: >550 Giga cells/L); neutrophil count (low: <1.5 Giga cells/L); white blood cell (WBC) count (low: <3 Giga cells/L and high: >20 Giga cells/L). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category. Participants were counted twice if the participant had both values that changed 'To Low' and 'To High'.
Time Frame: Up to Day 43
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 12 | 24
Participants
  Hematocrit, To Low | 0 | 0
  Hematocrit, To within range or no change | 12 | 24
  Hematocrit, To High | 0 | 0
  Hemoglobin, To Low | 0 | 0
  Hemoglobin, To within range or no change | 12 | 24
  Hemoglobin, To High | 0 | 0
  Lymphocytes, To Low | 1 | 0
  Lymphocytes, To within range or no change | 11 | 24
  Lymphocytes, To High | 0 | 0
  Platelet count, To Low | 0 | 0
  Platelet count, To within range or no change | 12 | 22
  Platelet count, To High | 0 | 2
  Neutrophil count, To Low | 0 | 1
  Neutrophil count, To within range or no change | 12 | 23
  Neutrophil count, To High | 0 | 0
  WBC, To Low | 0 | 2
  WBC To within range or no change | 12 | 24
  WBC, To High | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Worst Case Abnormal Hematology Parameters by PCI Criteria
Description: Hematology parameters with their PCI ranges were: hematocrit (high: >0.54 proportion of red blood cells in blood and low: change from BL<0.075); hemoglobin (high: >180 g/L and low: change from BL<25 g/L); lymphocytes (low: <0.8 Giga cells/L); platelet count (low: <100 Giga cells/L and high: >550 Giga cells/L); neutrophil count (low: <1.5 Giga cells/L); WBC count (low: <3 Giga cells/L and high: >20 Giga cells/L). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category. Participants were counted twice if the participant had both values that changed 'To Low' and 'To High'.
Time Frame: From Day 44 to Day 112
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK2982772 60 mg TID OL
Number analyzed (Participants) | 35
Participants
  Hematocrit, To Low | 0
  Hematocrit, To within range or no change | 35
  Hematocrit, To High | 0
  Hemoglobin, To Low | 0
  Hemoglobin, To within range or no change | 35
  Hemoglobin, To High | 0
  Lymphocytes, To Low | 1
  Lymphocytes, To within range or no change | 34
  Lymphocytes, To High | 0
  Platelet count, To Low | 0
  Platelet count, To within range or no change | 35
  Platelet count, To High | 0
  Neutrophil count, To Low | 0
  Neutrophil count, To within range or no change | 35
  Neutrophil count, To High | 0
  WBC, To Low | 1
  WBC To within range or no change | 34
  WBC, To High | 0

7. Primary Outcome: Part A: Number of Participants With Worst Case Abnormal Urinalysis Results by Dipstick Method
Description: Urine samples were collected for the assessment of following urine parameters by dipstick method: glucose, protein, blood and ketones. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine glucose, protein, blood and ketones can be read as negative (-), trace, 1+, 2+, 3+, 4+, 5+ indicating proportional concentrations in the urine sample. Number of participants with abnormal results were reported as 'increase to trace' or 'increase to 1+, 2+, 3+, 4+, 5+' relative to BL (Day 1) value. Participants whose value was unchanged (e.g., Trace to Trace), or whose value was decreased, were recorded in the 'No change or Decreased' category.
Time Frame: Up to Day 43
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 11 | 24
Participants
  Glucose, No change or decreased | 11 | 24
  Glucose, Increase to Trace | 0 | 0
  Glucose, Increase to 1+ | 0 | 0
  Glucose, Increase to 2+ | 0 | 0
  Glucose, Increase to 3+ | 0 | 0
  Glucose, Increase to 4+ | 0 | 0
  Glucose, Increase to 5+ | 0 | 0
  Ketones, No change or decreased | 10 | 16
  Ketones, Increase to Trace | 0 | 3
  Ketones, Increase to 1+ | 0 | 3
  Ketones, Increase to 2+ | 1 | 1
  Ketones, Increase to 3+ | 0 | 1
  Ketones, Increase to 4+ | 0 | 0
  Ketones, Increase to 5+ | 0 | 0
  Occult Blood, No change or decreased | 7 | 21
  Occult Blood, Increase to Trace, | 2 | 2
  Occult Blood, Increase to 1+ | 0 | 1
  Occult Blood, Increase to 2+ | 2 | 0
  Occult Blood, Increase to 3+ | 0 | 0
  Occult Blood, Increase to 4+ | 0 | 0
  Occult Blood, Increase to 5+ | 0 | 0
  Protein, No change or Decreased | 8 | 19
  Protein, Increase to Trace | 2 | 4
  Protein, Increase to 1+ | 1 | 1
  Protein, Increase to 2+ | 0 | 0
  Protein, Increase to 3+ | 0 | 0
  Protein, Increase to 4+ | 0 | 0
  Protein, Increase to 5+ | 0 | 0

8. Primary Outcome: Part B: Number of Participants With Worst Case Abnormal Urinalysis Results by Dipstick Method
Description: as for outcome 7
Time Frame: From Day 44 to Day 112
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK2982772 60 mg TID OL
Number analyzed (Participants) | 34
Participants
  Glucose, No change or Decreased | 34
  Glucose, Increase to Trace | 0
  Glucose, Increase to 1+ | 0
  Glucose, Increase to 2+ | 0
  Glucose, Increase to 3+ | 0
  Glucose, Increase to 4+ | 0
  Glucose, Increase to 5+ | 0
  Ketones, No change or Decrease | 21
  Ketones, Increase to Trace | 9
  Ketones, Increase to 1+ | 2
  Ketones, Increase to 2+ | 2
  Ketones, Increase to 3+ | 0
  Ketones, Increase to 4+ | 0
  Ketones, Increase to 5+ | 0
  Occult Blood, No change or Decreased | 30
  Occult Blood, Increase to Trace | 2
  Occult Blood, Increase to 1+ | 1
  Occult Blood, Increase to 2+ | 1
  Occult Blood, Increase to 3+ | 0
  Occult Blood, Increase to 4+ | 0
  Occult Blood, Increase to 5+ | 0
  Protein, No change or Decreased | 30
  Protein, Increase to Trace | 3
  Protein, Increase to 1+ | 1
  Protein, Increase to 2+ | 0
  Protein, Increase to 3+ | 0
  Protein, Increase to 4+ | 0
  Protein, Increase to 5+ | 0

9. Primary Outcome: Part A: Number of Participants With Worst Case Abnormal Blood Pressure Results by PCI Criteria
Description: Vital signs were measured in a semi-supine position after 5 minutes rest and included body temperature, systolic and diastolic blood pressure. The clinical concern range for vital signs were: systolic blood pressure (SBP) (low: <85 and high: >160 millimeters of mercury [mmHg]); diastolic blood pressure (DBP) (low: <45 and high: >100 mmHg). Participants were counted in the worst case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: Up to Day 43
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 12 | 24
Participants
  DBP, To Low | 0 | 0
  DBP, To within range or no change | 12 | 24
  DBP, To High | 0 | 0
  SBP, To Low | 0 | 0
  SBP, To within range or no change | 12 | 24
  SBP, To High | 0 | 0

10. Primary Outcome: Part B: Number of Participants With Worst Case Abnormal Blood Pressure Results by PCI Criteria
Description: Vital signs were measured in a semi-supine position after 5 minutes rest and included body temperature, systolic and diastolic blood pressure. The clinical concern range for vital signs were: SBP (low: <85 and high: >160 mmHg); DBP (low: <45 and high: >100 mmHg). Participants were counted in the worst case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: From Day 44 to Day 112
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK2982772 60 mg TID OL
Number analyzed (Participants) | 35
Participants
  DBP, To Low | 0
  DBP, To within range or no change | 34
  DBP, To High | 1
  SBP, To Low | 0
  SBP, To within range or no change | 33
  SBP, To High | 2

11. Primary Outcome: Part A: Number of Participants With Worst Case Abnormal Heart Rate (HR) Results by PCI Criteria
Description: Vital signs were measured in a semi-supine position after 5 minutes rest which included HR. The clinical concern range for HR (low <40 beats per min [bpm] and high >100 bpm). Participants were counted in the worst case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: Up to Day 43
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 12 | 24
Participants
  HR, To Low | 0 | 0
  HR, To within range or no change | 11 | 24
  HR, To High | 1 | 0

12. Primary Outcome: Part B: Number of Participants With Worst Case Abnormal HR Results by PCI Criteria
Description: Vital signs were measured in a semi-supine position after 5 minutes rest which included HR. The clinical concern range for HR (low <40 bpm and high >100 bpm). Participants were counted in the worst case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: From Day 44 to Day 112
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK2982772 60 mg TID OL
Number analyzed (Participants) | 35
Participants
  HR, To Low | 0
  HR, To within range or no change | 35
  HR, To High | 0

13. Primary Outcome: Part A: Number of Participants With Worst-case Abnormal Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were recorded with the participants in a supine position using an ECG machine. Number of participants with worst-case clinically significant and not clinically significant abnormal ECG findings have been presented. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 43
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 12 | 24
Participants
  Abnormal-not clinically significant | 5 | 11
  Abnormal-clinically significant | 0 | 0

14. Primary Outcome: Part B: Number of Participants With Worst-case Abnormal ECG Findings
Description: as for outcome 13
Time Frame: From Day 44 to Day 112
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK2982772 60 mg TID OL
Number analyzed (Participants) | 35
Participants
  Abnormal-not clinically significant | 18
  Abnormal-clinically significant | 1

15. Secondary Outcome: Part A: Percentage of Participants Who Achieved an Absolute Mayo Endoscopy Subscore of 0 or 1 at Day 43
Description: The Mayo scoring system was used to assess UC disease activity, scoring ranges from 0 to 12, calculated as sum of 4 sub-scores, higher scores indicating more severe disease. The 4 sub-scores are stool frequency (0=normal number of stools;1=1 to 2 stools/day more than normal;2=3 to 4 stools/day more than normal;3= >4 stools/day more than normal); rectal bleeding (0=no blood seen; 1=visible blood with stools less than half the time;2= visible blood with stool half the time or more;3=passing blood alone); findings at endoscopy (0=normal or inactive disease;1=mild disease [erythema,decreased vascular pattern,mild friability];2=moderate disease [marked erythema, lack of vascular pattern, friability, erosions];3=severe disease [spontaneous bleeding, ulceration]); and physician's global assessment (PGA) (0=normal;1=mild;2=moderate;3=severe). Number of participants with Mayo endoscopic sub-score of 0 or 1 are presented. (range=0 to 3, higher scores indicating more severe disease).
Time Frame: Day 43
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 11 | 24
Percentage of participants
  Mayo endoscopy sub-score =0 | 0 | 4
  Mayo endoscopy sub-score=1 | 0 | 8

16. Secondary Outcome: Part B: Percentage of Participants Who Achieved an Absolute Mayo Endoscopy Subscore of 0 or 1 at Day 85
Description: The Mayo scoring system was used to assess UC disease activity, scoring ranges from 0 to 12, calculated as sum of 4 sub-scores, higher scores indicating more severe disease. The 4 sub-scores are stool frequency (0=normal number of stools; 1=1 to 2 stools/day more than normal; 2=3 to 4 stools/day more than normal; 3= >4 stools/day more than normal); rectal bleeding (0=no blood seen; 1=visible blood with stools less than half the time; 2= visible blood with stool half the time or more; 3=passing blood alone); findings at endoscopy (0=normal or inactive disease; 1=mild disease [erythema, decreased vascular pattern, mild friability]; 2=moderate disease [marked erythema, lack of vascular pattern, friability, erosions]; 3=severe disease [spontaneous bleeding, ulceration]); and PGA (0=normal; 1=mild; 2=moderate; 3=severe). Number of participants with Mayo endoscopic sub-score of 0 or 1 are presented. (range=0 to 3, higher scores indicating more severe disease).
Time Frame: Day 85
Population: Safety Population. Only those participants with data available at the specified time points were analyzed. All participants in Part B received GSK2982772 60 mg in Part B (OL Phase), however they were split into 2 arms as randomized in Part A to allow statistical comparison of efficacy outcomes.
Measure: Number; unit: Percentage of participants
Groups:
- GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL: Eligible participants with UC, received GSK2982772 60 mg (given as 2 tablets of 30 mg) TID orally for 42 days (from Day 1 to 43) in Part A (double blind phase), followed by GSK2982772 60 mg (given as 2 tablets of 30 mg) TID orally for 42 days (from Day 44 to 85) in Part B (open label phase). There was no wash out period in between Part A and B. All participants were followed up until Day 112. 1 participant was randomized to receive BID regimen instead of TID regimen prior to protocol amendment; however, BID and TID are presented in the same arm because the PK profile is comparable for BID & TID regimen
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 9 | 22
Percentage of participants
  Mayo endoscopy sub-score =0 | 0 | 5
  Mayo endoscopy sub-score=1 | 11 | 9

17. Secondary Outcome: Part A: Change From Baseline in Ulcerative Colitis Endoscopic Index of Severity (UCEIS) Total Score
Description: UCEIS was used as an additional tool to assess disease activity based on 3 sub-scales: 'endoscopic vascular pattern, bleeding, erosions and ulcerations'. UCEIS total score was calculated by sum of all 3 sub-scale scores. Total score ranges from 0 to 8, with higher scores indicating more severe disease. Individual sub-scales were vascular pattern (0=Normal, 1=Patchy loss, 2=Obliterated); bleeding (0=None, 1=Mucosal, 2=Luminal mild, 3=Luminal severe); erosions and ulcerations (0=None, 1=Erosions, 2=Superficial ulcer, 3=Deep ulcer). BL is defined as the latest pre-dose assessment at Screening (within 30 days prior to Day 1). Change from BL was calculated as post-BL visit value minus BL value.
Time Frame: Baseline (screening - within 30 days prior to Day 1) and Day 43
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 11 | 24
Scores on scale | -0.24 (0.428) | -0.42 (0.289)
Statistical Analysis 1: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = -0.18, 95% CI 2-sided [-1.23 to 0.87] — Analysis performed using a Mixed Models Repeated Measures (MMRM) model, adjusting for the following covariates: treatment, visit, Baseline value, and the treatment by visit and baseline value by visit interactions

18. Secondary Outcome: Part B: Change From Baseline in Ulcerative Colitis Endoscopic Index of Severity (UCEIS) Total Score
Description: UCEIS was used as an additional tool to assess disease activity based on 3 sub-scales: 'endoscopic vascular pattern, bleeding, erosions and ulcerations'. UCEIS total score was calculated by sum of all 3 sub-scale scores. Total score ranges from 0 to 8, with higher scores indicating more severe disease. Individual sub-scales were vascular pattern (0=Normal, 1=Patchy loss, 2=Obliterated); bleeding (0=None, 1=Mucosal, 2=Luminal mild, 3=Luminal severe); erosions and ulcerations (0=None, 1=Erosions, 2=Superficial ulcer, 3=Deep ulcer). Baseline is defined as the latest pre-dose assessment at Screening (within 30 days prior to Day 1). Change from BL was calculated as post-BL visit value minus BL value.
Time Frame: Baseline (screening - within 30 days prior to Day 1) and Day 85
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles). All participants in Part B received GSK2982772 60 mg in Part B (OL Phase), however they were split into 2 arms as randomized in Part A to allow statistical comparison of efficacy outcomes.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 9 | 22
Scores on scale | -0.84 (0.495) | -0.82 (0.318)
Statistical Analysis 1: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Least Square Mean Difference = 0.02, 95% CI 2-sided [-1.18 to 1.22] — Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline value, and the treatment by visit and baseline value by visit interactions

19. Secondary Outcome: Part A: Change From Baseline in Mean C Reactive Protein (CRP)
Description: Blood samples were collected to measure CRP. BL is defined as the latest pre-dose assessment on Day 1. Change from BL is the value at indicated time point minus BL value.
Time Frame: Baseline (Day 1, pre-dose) and Days 15, 29, 43
Population: Safety population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Least Squares Mean (Standard Error); unit: Milligrams per liter
Groups:
- Part A: Placebo TID DB; Part A: GSK2982772 60 mg TID DB: Eligible participants with UC, received GSK2982772 60 mg (given as 2 tablets of 30 mg) TID orally for 42 days in Part A (double blind phase).
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 11 | 24
Milligrams per liter
  Day 15, n=11,24 | 0.25 (1.648) | 0.20 (1.112)
  Day 29, n=11, 23: number analyzed (Participants) | 11 | 23
  Day 29, n=11, 23 | 1.34 (1.119) | -1.84 (0.782)
  Day 43, n=11, 24 | 1.06 (1.854) | -0.64 (1.251)
Statistical Analysis 1: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = -0.05, 95% CI 2-sided [-4.11 to 4.02] — Day 15. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline value, and the treatment by visit and Baseline value by visit interactions
Statistical Analysis 2: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = -3.17, 95% CI 2-sided [-5.99 to -0.35] — Day 29. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline value, and the treatment by visit and Baseline value by visit interactions
Statistical Analysis 3: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = -1.69, 95% CI 2-sided [-6.26 to 2.88] — Day 43. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline value, and the treatment by visit and Baseline value by visit interactions

20. Secondary Outcome: Part B:Change From Baseline in Mean CRP
Description: as for outcome 19
Time Frame: Baseline (Day 1, pre-dose) and Days 57, 71, 85
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: Milligrams per liter
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 11 | 23
Milligrams per liter
  Day 57, n=11,23 | -2.61 (1.740) | -2.32 (1.186)
  Day 71, n=11, 22: number analyzed (Participants) | 11 | 22
  Day 71, n=11, 22 | -2.82 (1.510) | -2.71 (1.040)
  Day 85, n=10, 22: number analyzed (Participants) | 10 | 22
  Day 85, n=10, 22 | -2.77 (1.616) | -1.66 (1.092)
Statistical Analysis 1: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Least Square Mean Difference = 0.29, 95% CI 2-sided [-4.01 to 4.59] — Day 57. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline value, and the treatment by visit and Baseline value by visit interactions
Statistical Analysis 2: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Least Square Mean Difference = 0.11, 95% CI 2-sided [-3.64 to 3.85] — Day 71. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline value, and the treatment by visit and Baseline value by visit interactions
Statistical Analysis 3: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Least Square Mean Difference = 1.12, 95% CI 2-sided [-2.87 to 5.10] — Day 85. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline value, and the treatment by visit and Baseline value by visit interactions

21. Secondary Outcome: Part A: Change From Baseline in Fecal Calprotectin (FCP)
Description: Fecal sample were collected to measure FCP. BL is defined as the latest pre-dose assessment on Day 1. Change from BL is the value at indicated time point minus BL value.
Time Frame: Baseline (Day 1, pre-dose) and Days 15, 29, 43
Population: as for outcome 19
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Microgram per gram
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 11 | 23
Microgram per gram
  Day 15, n=10, 23: number analyzed (Participants) | 10 | 23
  Day 15, n=10, 23 | 0.78 (39.2) | 0.55 (25.1)
  Day 29, n=11, 23 | 1.23 (33.5) | 0.54 (22.3)
  Day 43, n=11, 22: number analyzed (Participants) | 11 | 22
  Day 43, n=11, 22 | 1.90 (40.7) | 0.44 (27.1)
Statistical Analysis 1: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Ratio = 0.70, 95% CI 2-sided [0.27 to 1.80] — Day 15. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, log-transformed Baseline value, and the treatment by visit and log-transformed baseline value by visit interactions
Statistical Analysis 2: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Ratio = 0.44, 95% CI 2-sided [0.20 to 1.00] — Day 29. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, log-transformed Baseline value, and the treatment by visit and log-transformed baseline value by visit interactions
Statistical Analysis 3: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Ratio = 0.23, 95% CI 2-sided [0.09 to 0.62] — Day 43. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, log-transformed Baseline value, and the treatment by visit and log-transformed baseline value by visit interactions

22. Secondary Outcome: Part B:Change From Baseline in FCP
Description: as for outcome 21
Time Frame: Baseline (Day 1, pre-dose) and Days 57, 71, 85
Population: as for outcome 18
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Microgram per gram
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 11 | 23
Microgram per gram
  Day 57, n=11, 23 | 1.13 (27.7) | 0.56 (18.7)
  Day 71, n=11, 22: number analyzed (Participants) | 11 | 22
  Day 71, n=11, 22 | 0.69 (42.1) | 0.39 (28.9)
  Day 85, n=11, 22: number analyzed (Participants) | 11 | 22
  Day 85, n=11, 22 | 0.48 (39.9) | 0.40 (27.2)
Statistical Analysis 1: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Ratio = 0.49, 95% CI 2-sided [0.25 to 0.97] — Day 57. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, log-transformed Baseline value, and the treatment by visit and log-transformed baseline value by visit interactions
Statistical Analysis 2: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Ratio = 0.56, 95% CI 2-sided [0.20 to 1.57] — Day 71. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, log-transformed Baseline value, and the treatment by visit and log-transformed baseline value by visit interactions
Statistical Analysis 3: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Ratio = 0.82, 95% CI 2-sided [0.31 to 2.18] — Day 85. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, log-transformed Baseline value, and the treatment by visit and log-transformed baseline value by visit interactions

23. Secondary Outcome: Part A: Change From Baseline in Modified Riley Scale Score (MRS)
Description: The MRS is a 4-point scale (none, mild, moderate and severe) which scores histologic activity based on localization and quantification of neutrophils in the mucosa. MRS Score ranges from 0 to 7, with higher scores indicates more severity. 0= Normal biopsy, 1= Lamina propria neutrophils only (Scattered individual neutrophils), 2= Lamina propria neutrophils only (Patchy collections of neutrophils), 3= Lamina propria neutrophils only (Diffuse neutrophils infiltrate), 4= Cryptitis/crypt abscesses (<25% crypts involved), 5= Cryptitis/crypt abscesses (25% to 74% crypts involved), 6= Cryptitis/crypt abscesses (>=75% crypts involved), 7= Erosion or ulceration present. Score 0 indicates normal condition; 1 to 3 indicates mild condition; 4 to 6 indicates moderate condition and score 7 indicates severe condition. BL is defined as the latest pre-dose assessment. Change from BL is the value at indicated time point minus BL value.
Time Frame: Baseline (Day 1, pre-dose) and Day 43
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 10 | 23
Scores on scale | 0.04 (0.842) | 0.04 (0.558)
Statistical Analysis 1: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = 0.01, 95% CI 2-sided [-2.05 to 2.07] — Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline score, and the treatment by visit and Baseline score by visit interactions

24. Secondary Outcome: Part B: Change From Baseline in MRS Score
Description: as for outcome 23
Time Frame: Baseline (Day 1, pre-dose) and Day 85
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 9 | 21
Scores on scale | -0.72 (0.894) | -0.65 (0.576)
Statistical Analysis 1: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Least Square Mean Difference = 0.08, 95% CI 2-sided [-2.11 to 2.27] — [estimate comment as in outcome 23, analysis 1]

25. Secondary Outcome: Part A: Change From Baseline in Geboes Index Total Score
Description: Geboes score is a 7-items instrument which classifies histologic changes and generates a score from 0 to 5.4. The 7 items are: grade 0=structural-architectural changes (scored from 0.0 to 0.3); grade 1=chronic inflammatory infiltrate (scored from 1.0 to 1.3); grade 2A=lamina propria neutrophils (scored from 2.0 to 2.3), grade 2B= lamina propria eosinophils (scored from 2.0 to 2.3); 3=neutrophils in the epithelium (scored from 3.0 to 3.3); 4=crypt destruction (scored from 4.0 to 4.3); 5=erosions or ulceration (scored from 5.0 to 5.4). The most severe observation that the histopathologist sees on the slide is considered as the Geboes index total score, ranges from 0 to 5.4, with higher scores indicates severe disease. BL is defined as the latest pre-dose assessment before Day 1. Change from BL is the value at indicated time point minus BL value.
Time Frame: Baseline and Day 43
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 10 | 23
Scores on scale | 1.04 (1.847) | 0.28 (1.223)
Statistical Analysis 1: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = -0.76, 95% CI 2-sided [-5.29 to 3.77] — [estimate comment as in outcome 23, analysis 1]

26. Secondary Outcome: Part B: Change From Baseline in Geboes Index Total Score
Description: as for outcome 25
Time Frame: Baseline and Day 85
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 9 | 21
Scores on scale | -0.67 (1.981) | -1.47 (1.286)
Statistical Analysis 1: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Least Square Mean Difference = -0.80, 95% CI 2-sided [-5.68 to 4.08] — [estimate comment as in outcome 23, analysis 1]

27. Secondary Outcome: Part A: Number of Participants Who Achieved Mayo Clinical Response
Description: Mayo Clinical Response is defined as a >=3 points or >=30% improvement from BL in Total Mayo Score, along with a decrease in the rectal bleeding sub-score of >= 1 point. The Mayo scoring system ranges from 0 to 12, calculated as sum of 4 sub-scores, higher scores indicating more severe disease. The 4 sub-scores are stool frequency (0=normal number of stools; 1=1 to 2 stools/day more than normal; 2=3 to 4 stools/day more than normal; 3= >4 stools/day more than normal); rectal bleeding (0=no blood seen; 1=visible blood with stools less than half the time; 2= visible blood with stool half the time or more; 3=passing blood alone); findings at endoscopy (0=normal or inactive disease; 1=mild disease [erythema, decreased vascular pattern, mild friability]; 2=moderate disease [marked erythema, lack of vascular pattern, friability, erosions]; 3=severe disease [spontaneous bleeding, ulceration]); and PGA (0=normal; 1=mild; 2=moderate; 3=severe).
Time Frame: Day 43
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 11 | 24
Participants | 4 | 9

28. Secondary Outcome: Part B: Number of Participants Who Achieved Mayo Clinical Response
Description: as for outcome 27
Time Frame: Day 85
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 9 | 22
Participants | 5 | 11

29. Secondary Outcome: Part A: Number of Participants Who Achieved Mayo Clinical Remission
Description: Mayo clinical remission is defined as total mayo score of 2 points or lower, with no individual subscore exceeding 1 point. The Mayo scoring system ranges from 0 to 12, calculated as sum of 4 sub-scores, higher scores indicating more severe disease. The 4 sub-scores are stool frequency (0=normal number of stools; 1=1 to 2 stools/day more than normal; 2=3 to 4 stools/day more than normal; 3= >4 stools/day more than normal); rectal bleeding (0=no blood seen; 1=visible blood with stools less than half the time; 2= visible blood with stool half the time or more; 3=passing blood alone); findings at endoscopy (0=normal or inactive disease; 1=mild disease [erythema, decreased vascular pattern, mild friability]; 2=moderate disease [marked erythema, lack of vascular pattern, friability, erosions]; 3=severe disease [spontaneous bleeding, ulceration]); and PGA (0=normal; 1=mild; 2=moderate; 3=severe).
Time Frame: Day 43
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 11 | 24
Participants | 0 | 0

30. Secondary Outcome: Part B: Number of Participants Who Achieved Mayo Clinical Remission
Description: as for outcome 29
Time Frame: Day 85
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 9 | 22
Participants | 1 | 2

31. Secondary Outcome: Part A: Change From Baseline in Partial Mayo Score
Description: Partial Mayo Score is defined as the total score of 3 domain subscores-stool frequency, rectal bleeding and PGA. Scoring ranges from 0 to 9, higher scores indicating more severe disease. The Mayo scoring system has 4 sub-scores: Stool frequency (0=normal number of stools; 1=1 to 2 stools/day more than normal; 2=3 to 4 stools/day more than normal; 3= >4 stools/day more than normal); rectal bleeding (0=no blood seen; 1=visible blood with stools less than half the time; 2= visible blood with stool half the time or more;3=passing blood alone); findings at endoscopy (0=normal or inactive disease;1=mild disease[erythema,decreased vascular pattern,mild friability];2=moderate disease[marked erythema,lack of vascular pattern,friability,erosions];3=severe disease [spontaneous bleeding,ulceration]);and PGA (0=normal; 1=mild; 2=moderate; 3=severe). Change from BL=post-BL value minus BL value (screening-within 30 days prior to Day 1).
Time Frame: Baseline (Screening - within 30 days prior to Day 1) and at Days 15, 29, 43
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 11 | 24
Scores on scale
  Day 15 | -0.68 (0.493) | -1.04 (0.333)
  Day 29: number analyzed (Participants) | 11 | 23
  Day 29 | -1.05 (0.480) | -1.16 (0.324)
  Day 43 | -1.30 (0.557) | -1.64 (0.376)
Statistical Analysis 1: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = -0.36, 95% CI 2-sided [-1.58 to 0.86] — Day 15. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline score, and the treatment by visit and Baseline score by visit interactions
Statistical Analysis 2: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = -0.10, 95% CI 2-sided [-1.29 to 1.08] — Day 29. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline score, and the treatment by visit and Baseline score by visit interactions
Statistical Analysis 3: Comparison: Part A: Placebo TID DB vs Part A: GSK2982772 60 mg TID DB; Test type: Other; Least Square Mean Difference = -0.34, 95% CI 2-sided [-1.72 to 1.04] — Day 43. Analysis performed using a MMRM model, adjusting for the following covariates: treatment, visit, Baseline score, and the treatment by visit and Baseline score by visit interactions

32. Secondary Outcome: Part B: Change From Baseline in Partial Mayo Score
Description: Partial Mayo Score defined as total score of 3 domain subscores-stool frequency, rectal bleeding and PGA, ranges from 0 to 9, higher score indicate more severe disease. It has 4 sub-scores: Stool frequency (0=normal number of stools; 1=1 to 2 stools/day more than normal; 2=3 to 4 stools/day more than normal; 3= >4 stools/day more than normal); rectal bleeding (0=no blood seen; 1=visible blood with stools less than half the time; 2= visible blood with stool half the time or more;3=passing blood alone); findings at endoscopy (0=normal or inactive disease;1=mild disease[erythema,decreased vascular pattern,mild friability];2=moderate disease[marked erythema,lack of vascular pattern, friability, erosions];3=severe disease [spontaneous bleeding,ulceration]);and PGA (0=normal, 3=severe). Change from BL=post-BL value minus BL value (screening-within 30 days prior to Day 1).
Time Frame: Baseline and Day 85
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 11 | 22
Scores on scale | -2.87 (0.728) | -2.93 (0.502)
Statistical Analysis 1: Comparison: Placebo TID DB /GSK2982772 60 mg TID OL vs GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL; Test type: Other; Least Square Mean Difference = -0.06, 95% CI 2-sided [-1.87 to 1.75] — [estimate comment as in outcome 23, analysis 1]

33. Secondary Outcome: Part A: Pre-dose Plasma Concentration of GSK2982772
Description: Pre-dose blood sample was collected on Day 43 for the measurement of plasma concentration of GSK2982772. PK Population is defined as the participants in the safety population who received an active dose and for whom a GSK2982772 pharmacokinetic sample was obtained and analyzed
Time Frame: Day 43
Population: PK Population. Participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter
Arm/Group | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 23
Nanogram/milliliter | 131.749 (214.9127)

34. Secondary Outcome: Part A: Post-dose Plasma Concentrations of GSK2982772
Description: Post-dose blood sample were collected on Days 1 and 43 at 1, 2, 4 and 6 hours for the measurement of plasma concentration of GSK2982772.
Time Frame: Days 1 and 43: 1, 2, 4 and 6 hours post dose
Population: PK Population. Participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter
Arm/Group | Part A: GSK2982772 60 mg TID DB
Number analyzed (Participants) | 23
Nanogram/milliliter
  Day 1, 1 hour | 674.588 (412.8928)
  Day 1, 2 hours | 772.043 (378.5145)
  Day 1, 4 hours | 474.248 (309.5524)
  Day 1, 6 hours | 481.304 (679.5678)
  Day 43, 1 hour | 918.926 (508.8658)
  Day 43, 2 hours | 851.391 (340.6479)
  Day 43, 4 hours | 472.132 (246.0718)
  Day 43, 6 hours | 278.039 (187.2142)

35. Secondary Outcome: Part B: Trough Concentrations of GSK2982772 on Day 85
Description: Blood samples were collected for the measurement of trough plasma concentration of GSK2982772 on Day 85.
Time Frame: Day 85
Population: PK Population. Only those participants with data available at the specified time points were analyzed. All participants in Part B received GSK2982772 60 mg in Part B (OL Phase), however they were split into 2 arms as randomized in Part A to compare trough concentrations.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter
Arm/Group | Placebo TID DB /GSK2982772 60 mg TID OL | GSK2982772 60 mg TID DB /GSK2982772 60 mg TID OL
Number analyzed (Participants) | 10 | 24
Nanogram/milliliter | 47.970 (78.9909) | 150.642 (305.3144)

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected from the start of study treatment (Day 1) up to Day 43 in Part A and from Day 44 till follow up visit (Day 112) in Part B.
Description: SAEs and Non-SAEs were reported for the Safety Population which comprised of all participants who received at least one dose of study treatment. Adverse events are presented treatment wise.
Arm/Group | Part A: Placebo TID DB | Part A: GSK2982772 60 mg TID DB | Part B: GSK2982772 60 mg TID OL
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/24 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/24 | 2/35
Other Adverse Events (participants affected / at risk) | 7/12 | 13/24 | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo TID DB (N=12) | Part A: GSK2982772 60 mg TID DB (N=24) | Part B: GSK2982772 60 mg TID OL (N=35)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo TID DB (N=12) | Part A: GSK2982772 60 mg TID DB (N=24) | Part B: GSK2982772 60 mg TID OL (N=35)
Headache (Nervous system disorders) | 1 (1) | 6 (10) | 6 (7)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT02903966/SAP_000.pdf
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02903966/Prot_001.pdf